CLINICAL TRIAL: NCT04837339
Title: Diagnostic and Prognostic Biomarkers of Transplant Dysfunction in the Context of Lung Transplantation
Acronym: DATACOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019_0015
Record Dates: First submitted 2020-11-02; First posted 2021-04-08 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Lung Transplant Rejection; Lung Transplant Failure; Lung Transplant; Complications; Lung Transplant Failure and Rejection
Keywords: DATACOL
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with lung disease requiring transplantation or who have undergone lung transplantation (Other): There is no intervention to be administered.
  Interventions: Other: Collection of biological samples

INTERVENTIONS:
Other: Collection of biological samples — Blood sample, biopsies sample, hair sample.

SUMMARY:
Transplant results vary considerably from one organ to another. Lung transplantation has poorer long-term outcomes than other solid organ transplants, with a current median post-transplant survival of 6.0 years. Allograft rejection remains the leading cause of morbidity and mortality in all organ groups and is the leading cause of death, accounting for more than 40% of deaths beyond the first year after lung transplantation.

Each dysfunctions impacts the fate of the graft and therefore the survival of the recipient. Their early and precise diagnosis is therefore a major issue. The identification of the pathophysiological mechanisms underlying these different subtypes of dysfunction (transcriptomics, polymorphism of target genes of the immune system or tissue repair, cell phenotyping) is an essential step. It can only be done on the basis of a collection of samples linked to a clinical database allowing to contextualize each sample.

ELIGIBILITY:
Inclusion Criteria:

* Men or women over 15 years of age
* Suffering from a lung condition requiring a transplant planned at Foch Hospital or being followed up at Foch Hospital following a lung transplant
* Have signed the informed consent form and for patients aged 15 to 18 years that the person(s) exercising parental authority has/have signed the informed consent.
* Be affiliated with a Health Insurance plan.

Exclusion Criteria:

* Pregnant, parturient and/or lactating woman
* Hemoglobin level less than or equal to 8g/dl
* Persons of full age who are subject to a legal protection measure or who are unable to express their consent
* Persons under the protection of justice
* Not being able to follow the study requirements for geographical, social or psychological reasons
* Patient refusal.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2022-03-17 (Actual); Primary Completion 2037-03 (Estimated); Study Completion 2037-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate non-invasive markers of dysfunction to stratify the risk of rejection, present in the blood during the first year after transplantation (blood immunomarkers). | 15 years
  Correlation between blood biomarkers (cell free DNA, Donor Specific Antibodies characterization) and graft rejection.

SECONDARY OUTCOMES:
Evaluate relevant gene sets associated with high or low risk profiles of acute dysfunction and rejection (intragraft expression). | 15 years
  Correlation of biomarkers (graft) with the functionality of the allograft
Stratify lung transplant recipients using non-invasive biomarkers and a gene expression profile for risk of allograft loss based on first year post-transplant data | 15 years
  Assessment of the risk of graft loss based on biomarker variations in repeated measurements.
Identify biomarkers and gene sets associated with response to immunosuppressive treatments of rejection | 15 years
  Correlation between gene expression in lung transplants and response to treatment of rejection
Evaluate the costs associated with the use of invasive and non-invasive strategies to define the risk of allograft rejection. | 15 years
  Costs incurred to define the risk of allograft rejection
Assessing patient acceptability and well-being using invasive and non-invasive biomarkers | 15 years
  Variation in patient well-being with the use of a non-invasive strategy to define the risk of allograft rejection

CONTACTS AND LOCATIONS:
Locations (1):
- Roux, Suresnes, France

IPD SHARING:
Plan to Share IPD: Undecided